CLINICAL TRIAL: NCT00941122
Title: Comparison of Elution Swab (ESwab) and Amies Transport Swabs for Screening Patients for Methicillin Resistant Staphylococcus Aureus (MRSA) and Vancomycin Resistant Enterococci (VRE) Colonization
Acronym: MRSA VRE
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Christine Lee, McMaster University
Organization: McMaster University (Other)
Other Study IDs: MRSA.VRE.Detection
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Eluted Swab
Keywords: MRSA, VRE

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRSA/VRE patients: patients known to be colonized with MRSA/VRE
  Interventions: Device: Eluted Swab

INTERVENTIONS:
Device: Eluted Swab — Comparison of Eluted Swab with AMIES swab for detection of MRSA/VRE

SUMMARY:
1.To assess whether the Elution swab (ESwab) is superior to Amies transport swabs for the detection of Methicillin Resistant Staphylococcus aureus (MRSA) and Vancomycin Resistant Enterococci (VRE) in colonized patients and to determine whether nasal cultures alone is sufficient for detection of MRSA isolates in hospitalized patients. 2.To assess patient comfort in the use of the ESwab vs. Amies Transport swab for screening patients for methicillin resistant Staphylococcus aureus and vancomycin-resistant Enterococcus.

DETAILED DESCRIPTION:
MRSA is a major cause of nosocomial and life threatening infections. Infections with MRSA have been associated with a significantly higher morbidity, mortality and costs than methicillin-susceptible S. aureus (MSSA).1 Selection of these organisms has been greatest in the healthcare setting; however, MRSA have also become more prevalent in the community.2 To control the transmission of MRSA, the Society for Healthcare Epidemiology of America (SHEA) has recommended guidelines, which include an active surveillance program to identify potential reservoirs and a rigorous infection control program to control the spread of MRSA. Accurate identification of patients colonized with MRSA is essential in managing the transmission of the organism. It is currently unknown whether the currently utilized collection rayon swab is the optimal swab in detecting colonized patients The purpose of this study is to directly compare whether Eluted (ESwab) swab is superior to the currently utilized rayon swab in identifying MRSA/VRE colonized patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitallized patients known to be colonized with MRSA/VRE

Exclusion Criteria:

* Unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients known to be colonized with MRSA/VRE
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
1. To assess whether the Elution swab (ESwab) is superior to Amies transport swabs for the detection of MRSA/VRE | 12 months
1. To assess whether the Elution swab (ESwab) is superior to Amies transport swabs for the detection of MRSA/VRE in colonized patients | 12 months

SECONDARY OUTCOMES:
To assess patient comfort in the use of the ESwab vs. Amies Transport swab for screening patients for methicillin resistant Staphylococcus aureus and vancomycin-resistant Enterococcus. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lee, MD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada